CLINICAL TRIAL: NCT06387589
Title: Effects of Static Stretching Versus Post Facilitation Stretch of Iliopsoas in Non-Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/5
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Stretching Group (Experimental): Core stabilization exercises along with Static Stretching of Iliopsoas (Hold for 7-8s x 10 reps) Week 1 Lifting the leg while lying in a prone position with the knee bent Week 2 Lifting the leg in a prone position with a straight knee Week 3 Stretch in the modified Thomas test position Week 4 Modified launch stretch
  Interventions: Procedure: Core stability exercises; Procedure: Static Stretching of Iliopsoas
- PFS Group (Experimental): Core stabilization exercises along with Post Facilitation Stretch of Iliopsoas (5-10s x 10 reps) Patient's position supine at the edge of the table, non-effected hip and knee in flexion, experimental thigh and leg hang on the edge of table. Extend the hip of the opposite thigh up to the barrier. After that, the patient flexes the hip against maximal resistance (isometric) and breathes in for 5-10 seconds. Tell the patient "Relax", whereas the therapist applies a rapid stretch to a new barrier and is held for 10 seconds.
  Interventions: Procedure: Core stability exercises; Procedure: Post Facilitation Stretch of Iliopsoas

INTERVENTIONS:
Procedure: Core stability exercises — Core stability Exercises will include:
  PLANK SIDE PLANK BIRD DOG MS GILL CURLUP PLANK + LEG RAISES SIDE PLANK + LEG RAISES PLANK + WALKS SIDE TO SIDE SIDE PLANK + TWIST BIRD DOG
Procedure: Static Stretching of Iliopsoas — Static Stretching of Iliopsoas (Hold for 7-8s x 10 reps) Week 1 Lifting the leg while lying in a prone position with the knee bent Week 2 Lifting the leg in a prone position with a straight knee Week 3 Stretch in the modified Thomas test position Week 4 Modified launch stretch
  Arms: Static Stretching Group
Procedure: Post Facilitation Stretch of Iliopsoas — Post Facilitation Stretch of Iliopsoas (5-10s x 10 reps) Patient's position supine at the edge of the table, non-effected hip and knee in flexion, experimental thigh and leg hang on the edge of table. Extend the hip of the opposite thigh up to the barrier. After that, the patient flexes the hip against maximal resistance (isometric) and breathes in for 5-10 seconds. Tell the patient "Relax", whereas the therapist applies a rapid stretch to a new barrier and is held for 10 seconds.
  Arms: PFS Group

SUMMARY:
This study is a randomized controlled trial and the purpose of this study is to determine the effects of Static Stretching Versus Post Facilitation Stretch of Iliopsoas combined with core stability exercises in Non-Specific Low Back Pain"

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of Static Stretching Versus Post Facilitation Stretch of Iliopsoas on Pain, physical function, lumbar ROM and Hip ROM in patients Non-Specific Low Back Pain" adults (age : 30-50 years )

1. Numeric pain rating scale
2. Goniometer
3. Inclinometer
4. Oswestry Disability Questionairre Data will be collected before and after the intervention protocol for each participant.

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post intervention scores will be recorded.

ELIGIBILITY:
Inclusion Criteria

* Gender: Both male and female
* Individuals aged 30-50 years
* Non-Specific low back pain for at least 3 months
* pain radiating no further than the buttock
* Pain range between 3-8 on NPRS
* Positive Thomas Test

Exclusion Criteria:

* Diagnosis of systemic metabolic and/or neurological disorder, neuromuscular disorders, pregnancy
* Patients who have been receiving any other physical therapy treatment for NSLBP in the same period of the interventions
* Patients having Low back pain with any specific cause

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  It will be measured using Numeric Pain Rating Scale.It has a scale of 0-10 or 0-100 points and can be given verbally or in writing.
Level of disability | 4 weeks
  It will be measured using Oswestry disability Index Questionairre
Lumbar Range of motion | 4 weeks
  Lumbar ROM will be measured using Inclinometer
Hip Range of motion | 4 Weeks
  Hip ROM will be measured using Goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan